CLINICAL TRIAL: NCT06402942
Title: Gamified Occupational Therapy for Adolescents With Duchenne Muscular Dystrophy
Acronym: DMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başak Çağla Arslan (Other Government)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Başak Çağla Arslan, Lecturer, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LHU20241004; LHÜ (Other: LHÜ)
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy; Gamification; Occupational Therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Gamified occupational therapy programme group
  Interventions: Other: Gamified occupational therapy programme
- Control group (Other): Classic occupational therapy group
  Interventions: Other: Classic occupational therapy programme

INTERVENTIONS:
Other: Gamified occupational therapy programme — Gamified occupational therapy program for the experimental group and classical occupational therapy program for the control group, which will be applied to both groups for eight weeks
  Arms: Experimental group
Other: Classic occupational therapy programme — Gamified occupational therapy program for the experimental group and classical occupational therapy program for the control group, which will be applied to both groups for eight weeks
  Arms: Control group

SUMMARY:
This research aims to improve the quality of life, occupational performance, occupational satisfaction and emotional health of young people with Duchenne muscular dystrophy compared to the classical occupational therapy program. The findings are planned to shed light on the development of new and effective strategies in the rehabilitation of adolescents with Duchenne muscular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Duchenne muscular dystrophy
* To be literate in Turkish
* To have scored 27 points or more on the Modified Mini Mental Test
* Having a computer, tablet and internet connection
* Volunteering to participate in the study by their parents and reading and signing the informed consent form

Exclusion Criteria:

* Having a neurological disease other than Duchenne muscular dystrophy and/or another diagnosed neurological disease accompanying Duchenne muscular dystrophy
* Having a cooperation problem that prevents completing the assessments for any reason
* Difficulty understanding and speaking the Turkish language

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Duchenne muscular dystrophy occurs mostly in boys and very rarely in girls. Girls are usually carriers.
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | At the start of the evaluations
Modified Mini Mental State Test | before and after the eight-week intervention programs
Vignos lower extremity functional scale | before and after the eight-week intervention programs
  This scale was developed to assess the level of ambulation in neuromuscular diseases and consists of 10 stages. In this scale, the ambulation level of the person decreases from the first stage to the tenth stage.
Brooke upper extremity functional classification scale | before and after the eight-week intervention programs
  This scale was developed to assess the functional levels of the upper extremity in neuromuscular diseases and consists of 6 stages. In this scale, progression from the first stage to the sixth stage indicates a decrease in the functionality of the upper extremity.
The Pediatric Quality of Life Inventory 3.0 Neuromuscular Module | before and after the eight-week intervention programs
Canadian Occupational Performance Measure | before and after the eight-week intervention programs
Children's Depression Inventory | before and after the eight-week intervention programs
  Consisting of 27 items and using a 3-point Likert-type scale, this scale assesses the depression levels of children between the ages of 6-17. The total score of the scale, which measures the emotional state in the last 2 weeks, is 54 and the severity of depression increases as the total score increases. The cut-off value of the scale was determined as 19 points.
The Pediatric Quality of Life Inventory Multidimensional Fatigue Scale | before and after the eight-week intervention programs
  This scale consists of 18 items and 3 subsections: general fatigue (6 items), fatigue during sleep/rest (6 items) and cognitive fatigue (6 items). Separate scores can be calculated for each subsection and the total score is obtained by summing the scores obtained from these sections. High scores indicate low fatigue.
The Numeric Rating Scale - Pain | before and after the eight-week intervention programs
  This scale uses a 10-centimeter line. The left beginning of the line represents "no pain" (0 points) and the end of the line represents "excruciating pain" (10 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No